CLINICAL TRIAL: NCT02462525
Title: A Multicenter, Phase 1/1b, Open-Label, Dose-Escalation Study of ABBV-838, an Antibody Drug Conjugate, in Subjects With Relapsed and Refractory Multiple Myeloma
Brief Title: Dose-Escalation Study of ABBV-838, an Antibody Drug Conjugate, in Subjects With Relapsed and Refractory Multiple Myeloma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: No Go decision for ABBV-838
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M14-467; 2014-002609-39 (EudraCT Number)
Record Dates: First submitted 2015-05-26; First posted 2015-06-04 (Estimated); Last update posted 2018-09-13 (Actual); Status verified 2018-09

CONDITIONS: Multiple Myeloma
Keywords: relapsed multiple myeloma; antibody drug conjugate; refractory multiple myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — pomalidomide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ABBV-838 dose escalation (Experimental): Varying doses of ABBV-838
  Interventions: Drug: ABBV-838
- ABBV-838 plus pomalidomide/dexamethasone (Experimental): ABBV-838 to be evaluated with pomalidomide/dexamethasone.
  Interventions: Drug: ABBV-838; Drug: Pomalidomide; Drug: Dexamethasone

INTERVENTIONS:
Drug: ABBV-838 — Varying doses of ABBV-838
Drug: Pomalidomide — Administered orally per the label.
  Arms: ABBV-838 plus pomalidomide/dexamethasone
Drug: Dexamethasone — Administered orally per the label.
  Arms: ABBV-838 plus pomalidomide/dexamethasone

SUMMARY:
This is a Phase 1/1b, open-label, dose-escalation study designed to evaluate the safety, pharmacokinetics, and to determine the recommended Phase 2 dose of ABBV-838 in subjects with relapsed and refractory multiple myeloma.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group Performance Status of 0 to 2
* Not eligible for stem cell/bone marrow transplant or have refused stem cell/bone marrow transplant or have relapsed after autologous or allogeneic stem cell/bone marrow transplant
* Eligible for and agree to BM aspirate prior to treatment start
* Measurable disease M component in serum (≥ 0.5 g/dL) and/or urine (≥ 0.2 g excreted in a 24 hour collection sample)
* Must have received at least 3 prior lines of therapy including a proteasome inhibitor and an immunomodulatory agent or those who are double refractory to a PI and an immunomodulatory agent and have demonstrated disease progression (DP) on or within 60 days of completion of the last therapy; participants previously treated with an alkylating agent, in addition to an IMiD or proteasome inhibitor, are allowed to enroll in the trial
* Participants must have adequate liver, kidney, and bone morrow function
* Participants with a history of chronic heart failure must have cardiac ECHO indicating left ventricular ejection fraction (LVEF) ≥ 45% within 21 days prior to first dose of study drug
* Participants in the combination therapy arms must be eligible to receive pomalidomide/dexamethasone, bortezomib/dexamethasone or lenalidomide/dexamethasone or other approved agents per current prescribing information for MM.
* Participants who will receive combination therapy with Pomalidomide/Dexamethasone must have received at least two prior therapies including lenalidomide and a proteasome inhibitor and have demonstrated disease progression on or within 60 days of completion of the last therapy

Exclusion Criteria:

* Received anti-cancer therapy including chemotherapy, immunotherapy, radiation, biologic, any investigational therapy or herbal therapy within a period of 21 days prior to the first dose of ABBV-838, and have unresolved toxicities ≥ grade 2
* Concurrent metastatic solid tumors
* Non-Measurable M Protein (serum or urine) and measurable sFLC (< 100 mg/mL)
* Major surgery within 21 days prior to the first dose of ABBV-838
* Clinically significant uncontrolled condition(s) including but not limited to the following:

Grade ≥ 3 peripheral neuropathy or grade 2 peripheral neuropathy with pain Uncontrolled hypercalcemia Active uncontrolled infection Symptomatic congestive heart failure Unstable angina pectoris or cardiac arrhythmia Psychiatric illness/social situation that would limit compliance with the study

* Major immunologic reaction to any IgG containing agent or auristatin based agent
* Participants who are taking strong CYP3A4 inhibitors
* Positive for HIV (Human Immunodeficiency Virus) or with active hepatitis B and/or C
* Corneal pathology that would limit evaluation of loss in visual acuity associated with corneal deposits.
* Prior exposure to pomalidomide for subjects enrolling in the pomalidomide/dexamethasone combination arm.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2015-05-06 (Actual); Primary Completion 2017-12-06 (Actual); Study Completion 2017-12-06 (Actual)

PRIMARY OUTCOMES:
Maximum plasma concentration (Cmax) of ABBV-838 | Cycle 1 Day 1 (C1D1) and C3D1 pre- and post-dose; C1D4, C1D8, C1D15, C2D1, C2D15, C3D4, C3D8, C3D15, C4D1, and all subsequent ABBV-838 pre-dose dosing cycles
  The maximum plasma concentration (Cmax: measured in ng/ml) is the highest concentration that a drug achieves in the blood after the first dose, but before administration of a second dose.
Maximum tolerated dose of ABBV-838 | Up to 2 years from first dose of study
  The highest dose level at which less than 2 of 6 subjects or less than 33% of (if cohort is expanded beyond 6) subjects experience a dose limiting toxicity.

SECONDARY OUTCOMES:
Preliminary activity of ABBV-838 monotherapy | At screening, Cycle 1 Day 15 (C1D15), C3D15, C4D1, and for subjects who have been on ABBV-838 for ≥ 6 cycles, radiologic tumor assessments may be performed every 3 cycles per Investigator discretion up to approximately 3 years
  Response evaluation will be based on International Myeloma Working Group (IMWG) Response Criteria.

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie
Locations (19):
- United States (5):
  - The University of Chicago Medical Center /ID# 139403, Chicago, Illinois
  - University of Michigan Medical Center /ID# 139402, Ann Arbor, Michigan
  - Washington University School of Medicine /ID# 135708, St Louis, Missouri
  - Mount Sinai Medical Center /ID# 133569, New York, New York
  - The Sarah Cannon Research Institute /ID# 135814, Nashville, Tennessee
- France (3):
  - CHRU de Lille, Hopital Claude Huriez /ID# 133634, Lille
  - CHU de Nantes, Hotel Dieu - HME /ID# 133633, Nantes
  - CHU de la miletrie, Centre d'investigation clinique /ID# 147542, Poitiers
- Germany (6):
  - Universitaetsklinikum Koeln /ID# 141535, Cologne
  - Universitaetklinikum Dresden /ID# 141860, Dresden
  - Universitaetsklinikum Heidelberg /ID# 140046, Heidelberg
  - Universitaetsklinikum Schleswig-Holstein /ID# 141534, Kiel
  - Universitaetsklinikum Tuebingen /ID# 141074, Tübingen
  - Universitaetsklinikum Wuerzburg /ID# 141533, Würzburg
- Spain (5):
  - Hospital Clinic de Barcelona /ID# 141643, Barcelona
  - Hospital Universitario de la Princesa /ID# 140881, Madrid
  - Hospital Universitario 12 de Octubre /ID# 140878, Madrid
  - Clinica Universitaria de Navarra /ID# 141411, Pamplona-Navarra
  - Hospital Clinico Universitario Salamanca /ID# 140880, Salamanca

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Vij R, Nath R, Afar DEH, Mateos MV, Berdeja JG, Raab MS, Guenther A, Martinez-Lopez J, Jakubowiak AJ, Leleu X, Weisel K, Wong S, Gulbranson S, Sheridan JP, Reddy A, Paiva B, Singhal A, San-Miguel JF, Moreau P. First-in-Human Phase I Study of ABBV-838, an Antibody-Drug Conjugate Targeting SLAMF7/CS1 in Patients with Relapsed and Refractory Multiple Myeloma. Clin Cancer Res. 2020 May 15;26(10):2308-2317. doi: 10.1158/1078-0432.CCR-19-1431. Epub 2020 Jan 22. PMID 31969330